CLINICAL TRIAL: NCT07223073
Title: A Randomized Single-center, Double-blind, Two-cell Parallel-group Clinical Study Conducted in the Bangkok, Thailand Area, to Investigate the Clinical Efficacy of a New Toothpaste Containing 0.454% Stannous Fluoride as Compared to a Regular Fluoride Toothpaste Containing 0.76% Sodium Monofluorophosphate in Controlling Oral Malodor 12 Hours Post-brushing Overnight After 3 Weeks of Twice a Day (Morning and Evening) Product Use.
Brief Title: A Clinical Study Conducted in the Bangkok, Thailand Area, to Investigate the Clinical Efficacy of a New Toothpaste
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CRO-2017-10-OM-SNHW-THA-YPZ
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Oral Malodor
MeSH Terms: interventions — Tin Fluorides; fluorophosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Test 1 toothpaste (Experimental)
  Interventions: Drug: 0.454% stannous fluoride
- Test 2 Toothpaste (Active Comparator)
  Interventions: Drug: 0.76% sodium monofluorophosphate

INTERVENTIONS:
Drug: 0.454% stannous fluoride — fluoride toothpaste
  Arms: Test 1 toothpaste
Drug: 0.76% sodium monofluorophosphate — regular fluoride toothpaste
  Arms: Test 2 Toothpaste

SUMMARY:
To investigate the clinical efficacy of a new toothpaste containing 0.454% stannous fluoride as compared to a regular fluoride toothpaste containing 0.76% sodium monofluorophosphate on oral malodor reduction via organoleptic scores 12 hours post-brushing overnight after 3 weeks of twice a day (morning and evening) product use.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults between the ages of 18-70 (inclusive)
* Subjects must be in general good health
* Subjects must be in good oral health based on self-assessment
* Subjects must be available for the duration of the study for all time point assessments
* Subjects were required to possess a minimum of 20 natural uncrowned teeth (excluding third molars)
* Subjects were required to sign an Informed Consent form
* No known history or allergies to personal care/consumer products or their ingredients.

Exclusion Criteria:

* Participated in any other oral clinical studies during the duration of this study
* Had full or partial (upper or lower) dentures
* Women who are pregnant or lactating (breast feeding)
* Use of tobacco products, (5) History of allergies to common mouthwash ingredients
* Use of phenolic flavored products, such as mint flavored candies and chewing gum the morning of the study of during the sampling periods
* Immune compromised individuals (HIV, AIDS, immune suppressive drug therapy
* Individuals who, due to medical conditions cannot go without eating or drinking for the post use treatment evaluation time points (6-hours plus overnight).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

PRIMARY OUTCOMES:
Mean Organoleptic scores for each treatment group | Baseline, 12 hours post brushing and 3 weeks
  For each subject at each evaluation time point, the hedonic breath-odor scores assigned by the four (4) judges were averaged to yield a single subject-wise score. Statistical analyses were performed on these average organoleptic hedonic scores.

CONTACTS AND LOCATIONS:
Overall Officials: Terdphong Triratana, DDS, Principal Investigator — Mahidol University
Locations (1):
- M U International Oral Science Research, Ltd., Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No